CLINICAL TRIAL: NCT06599567
Title: THE EFFECT OF GRADED MOTOR IMAGERY AND NINTENDO WII-BASED BIOFEEDBACK TECHNIQUES ON ROTATOR CUFF PATHOLOGIES
Brief Title: Graded Motor Imagery and Biofeedback in Rotator Cuff Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Cansu ERCAN, Principal Investigator, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 8Z3KqXp1
Record Dates: First submitted 2024-09-12; First posted 2024-09-19 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Rotator Cuff Injuries; Rotator Cuff Injury; Rotator Cuff Syndrome
Keywords: graded motor imagery; pain; shoulder joint; rehabilitation; rotator cuff injuries
MeSH Terms: conditions — Rotator Cuff Injuries; Pain

STUDY DESIGN:
Intervention Model Description: 1. st group traditional therapy
  2. nd group : traditional therapy and graded motor imagery
  3. rd group traditional therapy and biofeedback training with nintendo wii
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Patients will not know which group they belong to and the physiotherapist who makes the evaluations will not know which treatment the patients receive. Our study will be conducted in a double-blind manner.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Traditional therapy (Active Comparator): Cold - Hot pack applications, TENS device application, which is a pain-relieving electrotherapy agent, therapeutic exercises
  Interventions: Other: Traditional therapy
- Graded motor imagery (Active Comparator): Cold-Hot pack applications, TENS device application, which is a pain-relieving electrotherapy agent, therapeutic exercises, graded motor imagery training (body right-left discrimination exercise, imagining the movement and exercising the opposite limb in front of the mirror).
  Interventions: Other: Graded motor imagery
- Nintendo Wİİ (Active Comparator): Cold - Hot pack applications, TENS device application, which is a pain-relieving electrotherapy agent, therapeutic exercises, games involving your relevant shoulder such as boxing and bowling on the Nintendo Wii game console.
  Interventions: Other: Nintendo Wİİ

INTERVENTIONS:
Other: Traditional therapy — Cold - Hot pack applications, TENS device application, which is a pain-relieving electrotherapy agent, therapeutic exercises
  Arms: Traditional therapy
Other: Graded motor imagery — Cold-Hot pack applications, TENS device application, which is a pain-relieving electrotherapy agent, therapeutic exercises, graded motor imagery training (body right-left discrimination exercise, imagining the movement and exercising the opposite limb in front of the mirror).
  Arms: Graded motor imagery
Other: Nintendo Wİİ — Cold - Hot pack applications, TENS device application, which is a pain-relieving electrotherapy agent, therapeutic exercises, games involving your relevant shoulder such as boxing and bowling on the Nintendo Wii game console.
  Arms: Nintendo Wİİ

SUMMARY:
Purpose: This study aims to compare the effectiveness of conventional therapy, Graded Motor Imagery (GMI), and Nintendo Wii-based biofeedback therapy in patients with rotator cuff injuries. The goal is to evaluate the impact of these three methods on pain management, range of motion (ROM), patient satisfaction, and functional performance.

Hypotheses:

There is no significant difference in pain management between conventional therapy, GMI, and Wii-based biofeedback therapy.

There is no significant difference in shoulder ROM between the three therapies. There is no significant difference in patient satisfaction among the therapies. There is no significant difference in functional performance improvement between the therapies.

Methods: A randomized, double-blind, controlled trial will be conducted with 36 patients with rotator cuff injuries. They will be randomly assigned to one of three groups and undergo 6 weeks of treatment. Pain, ROM, and functional performance will be assessed pre- and post-treatment. Data will be analyzed using ANOVA.

Potential Outcomes/Significance: The study may show that innovative approaches like GMI and Wii-based biofeedback therapy are effective treatment options. Results could contribute to developing new strategies for treating chronic pain and motor dysfunctions.

DETAILED DESCRIPTION:
Study Title: Comparative Effectiveness of Conventional Therapy, Graded Motor Imagery (GMI), and Nintendo Wii-Based Biofeedback Therapy in Rotator Cuff Injuries

Purpose: The primary aim of this study is to compare the effectiveness of three different therapeutic interventions-conventional therapy, Graded Motor Imagery (GMI), and Nintendo Wii-based biofeedback therapy-in managing rotator cuff injuries. The study will evaluate the impact of these therapies on key outcomes including pain management, shoulder range of motion (ROM), patient satisfaction, and functional performance. By comparing these methods, the study seeks to determine which therapy offers the best overall benefit for patients with rotator cuff injuries.

Hypotheses:

Hypothesis 1: There is no significant difference in pain management between conventional therapy, GMI, and Wii-based biofeedback therapy.

Alternative Hypothesis (H1): Significant differences in pain management exist among these therapies.

Hypothesis 2: There is no significant difference in shoulder ROM between conventional therapy, GMI, and Wii-based biofeedback therapy.

Alternative Hypothesis (H1): Significant differences in shoulder ROM exist among these therapies.

Hypothesis 3: There is no significant difference in patient satisfaction among conventional therapy, GMI, and Wii-based biofeedback therapy.

Alternative Hypothesis (H1): Significant differences in patient satisfaction exist among these therapies.

Hypothesis 4: There is no significant difference in functional performance improvement between conventional therapy, GMI, and Wii-based biofeedback therapy.

Alternative Hypothesis (H1): Significant differences in functional performance improvement exist among these therapies.

Methods: This study will use a randomized, double-blind, controlled trial design. A total of 36 patients diagnosed with rotator cuff injuries will be randomly assigned to one of three treatment groups: conventional therapy, Graded Motor Imagery (GMI), or Nintendo Wii-based biofeedback therapy. Each group will undergo their respective treatment for a duration of 6 weeks. The effectiveness of each treatment will be assessed through measurements taken before and after the intervention. Pain levels, shoulder ROM, and functional performance will be evaluated using standardized assessment tools. Statistical analysis will be performed using ANOVA to compare outcomes across the three treatment groups.

Potential Outcomes/Significance: The results of this study have the potential to highlight the effectiveness of innovative therapies like GMI and Wii-based biofeedback therapy in the treatment of rotator cuff injuries. If these methods are found to be more effective than conventional therapy, they could represent valuable additions to treatment options for patients suffering from chronic pain and motor dysfunctions. The findings may contribute to the development of new, evidence-based strategies for managing rotator cuff injuries and improving patient outcomes in rehabilitation settings.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18-65
* A rotator cuff injury was diagnosed and conservative treatment was decided
* Volunteer for research
* People who can read, write and understand Turkish

Exclusion Criteria:

* Having neurological findings of cervical origin
* An additional different orthopedic problem in the same shoulder (Full thickness rotator cuff tear, adhesive capsulitis and glenohumeral instability)
* Uncooperative or mental problem
* Neurological, vascular and cardiac problem that limits function

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2024-09-25 (Actual); Primary Completion 2025-05-25 (Actual); Study Completion 2025-05-25 (Actual)

PRIMARY OUTCOMES:
quickDASH short form | From enrollment to the end of treatment at 6 weeks
  QuickDASH will be used to assess upper extremity functional limitations and symptoms in patients with rotator cuff injuries Scoring: QuickDASH consists of 11 questions, each rated on a scale from 1 to 5. The final score is calculated between 0 (no difficulty) and 100 (extreme difficulty)

SECONDARY OUTCOMES:
Shoulder Pain | From enrollment to the end of treatment at 6 weeks
  NPRS (Numeric Pain Rating Scale) is a self-reported scale used to assess the intensity of pain. If you are conducting research on shoulder and arm injuries, such as rotator cuff pathologies, you can use this scale to evaluate the patients' pain levels.
  NPRS is an 11-point scale where the patient rates their pain from 0 (no pain) to 10 (worst possible pain)
Range of motion | From enrollment to the end of treatment at 6 weeks
  ROM (Range of Motion) is an objective measurement used to assess the mobility and flexibility of joints. If you are conducting research on shoulder injuries such as rotator cuff pathologies, you can use ROM assessments to evaluate improvements in joint mobility.
  ROM is usually measured in degrees using a goniometer. Specific movements like shoulder flexion, extension, abduction, and rotation are assessed.
Kinesiophobia | From enrollment to the end of treatment at 6 weeks
  The Tampa Scale of Kinesiophobia (TSK) is a self-reported questionnaire used to assess the fear of movement or re-injury in patients. If you are conducting research on shoulder injuries such as rotator cuff pathologies, you can use this scale to evaluate patients' fear of movement and its impact on recovery.
  The TSK consists of 17 items, each rated on a 4-point Likert scale. The total score ranges from 17 to 68, with higher scores indicating greater fear of movement.
Global Rating of Change | From enrollment to the end of treatment at 6 weeks
  The Global Rating of Change (GRC) is a self-reported scale used to measure a patient's perception of overall improvement or deterioration over time. If you are conducting research on rotator cuff injuries, you can use the GRC to evaluate patients' subjective assessment of their progress.
  The GRC is typically measured on a scale ranging from -5 (a very great deal worse) to +5 (a very great deal better), with 0 indicating no change.
Lateralization | From enrollment to the end of treatment at 6 weeks
  The Recognise app is a tool used to assess lateralization, which involves identifying left and right body parts to measure motor imagery and cortical representation. If you are conducting research on rotator cuff injuries, you can use this app to evaluate patients' ability to recognize and distinguish between left and right body parts, which can be important in assessing changes in cortical representation and motor imagery.

CONTACTS AND LOCATIONS:
Overall Officials: Cansu Ercan, Principal Investigator — Unaffiliated&amp;amp;amp;amp;amp;amp;#34;
Locations (1):
- Istanbul University- Cerrahpaşa, Istanbul, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD, all IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: November 2024 - November 2025
Access Criteria: Healthcare professionals doing research in this field

REFERENCES:
- [Background] Suso-Marti L, La Touche R, Angulo-Diaz-Parreno S, Cuenca-Martinez F. Effectiveness of motor imagery and action observation training on musculoskeletal pain intensity: A systematic review and meta-analysis. Eur J Pain. 2020 May;24(5):886-901. doi: 10.1002/ejp.1540. Epub 2020 Feb 20. PMID 32031724
- [Background] Hoyek N, Di Rienzo F, Collet C, Hoyek F, Guillot A. The therapeutic role of motor imagery on the functional rehabilitation of a stage II shoulder impingement syndrome. Disabil Rehabil. 2014;36(13):1113-9. doi: 10.3109/09638288.2013.833309. Epub 2014 Feb 28. PMID 24575717
- See also: The therapeutic role of motor imagery on the functional rehabilitation of a stage II shoulder impingement syndrome — https://pubmed.ncbi.nlm.nih.gov/24575717/
- See also: Effectiveness of motor imagery and action observation training on musculoskeletal pain intensity: A systematic review and meta-analysis — https://pubmed.ncbi.nlm.nih.gov/32031724/
- Available data/document: Individual Participant Data Set: sample size — https://bmjopen.bmj.com/content/10/11/e039976 — reference article to see sample size with g power
- Available data/document: Study Protocol: Nintendo Wii protocol — https://pubmed.ncbi.nlm.nih.gov/28330586/
- Available data/document: Study Protocol: Graded motor imagery protocol — https://pubmed.ncbi.nlm.nih.gov/32003812/